CLINICAL TRIAL: NCT02916420
Title: A Multicenter, Single-arm, Open-label Study to Evaluate the Efficacy and Safety of Pomalidomide in Combination With Low-dose Dexamethasone in Chinese Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Efficacy and Safety of Pomalidomide in Combination With Low-dose Dexamethasone in Chinese Patients With Relapsed and Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-135-Ⅲ
Record Dates: First submitted 2016-09-24; First posted 2016-09-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Pomalidomide plus low-dose Dexamethasone
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — 4mg/day, d1-d21, 28 days per cycle
Drug: Dexamethasone — ≤70 years,40mg/day; >70 years,20mg/day, d1、d8、d15、d22, 28 days per cycle

SUMMARY:
This study aims to assess the efficacy and safety of pomalidomide in combination with low-dose dexamethasone in Chinese patients with relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of multiple myeloma
* Subjects must have received at least 2 prior therapies. Subjects must have undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of bortezomib (either in separate regimens or within the same regimen). Subjects must also have documented evidence of progressive disease(PD) during or within 60 days (measured from the end of the last cycle) of completing treatment with the last anti-myeloma drug regimen used just prior to study entry.
* Subjects must have measurable disease: serum M-protein ≥ 5 g/L or urine M-protein ≥ 200 mg/24 hours or the involved free light chain being ≥100 mg/L when serum free light chain ratio (κ/λ ratio < 0.26 or > 1.65) is abnormal
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤2
* Life expectancy >3 months
* For female patients,

  * naturally postmenopausal for at least 24 months, or take surgical sterilization
  * Women of childbearing potential must:

    1. have 2 negative pregnancy tests before initiating pomalidomide. The first test should be performed within 10-14 days, and the second test within 24 hours prior to initiating pomalidomide
    2. commit either to abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control, beginning 4 weeks prior to initiating pomalidomide treatment, during therapy, and continuing for 4 weeks following discontinuation of pomalidomide therapy
    3. agree to perform the pregnancy testing during the study
* Male patients must always use a condom during any sexual contact with females of reproductive potential while taking pomalidomide and for up to 4 weeks after discontinuing pomalidomide, even if they have undergone a successful vasectomy. Meanwhile male patients taking pomalidomide must not donate sperm.
* Subjects agree not to share medication with another person
* Subjects are able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Any serious medical conditions, laboratory abnormality, or psychiatric illness that would prevent the patient from complying to the protocol or put the patient's safety at risk
* Evidence of uncontrolled cardiovascular disease, such as congestive heart failure, unstable angina, myocardial infarction within 12 months prior to enrollment
* Any of the following laboratory abnormalities:

  * ANC < 1×10^9/L
  * PLT < 75×10^9/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; or PLT < 30×10^9/L for subjects in whom ≥50% of bone marrow nucleated cells are plasma cells
  * Creatinine Clearance < 45 mL/min
  * AST or ALT > 3.0 x ULN
  * Serum total bilirubin > 34.2 μmol/L
  * Corrected serum calcium > 3.5 mmol/L
  * Hemoglobin < 80g/L
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following:

  * Basal or Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix or breast
  * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
* Serious, uncontrolled medical conditions or active infection, including but not limited to HIV antibody positive, HBsAg positive and HBV DNA copies > 1 × 10^3, hepatitis C virus antibody positive, uncontrolled diabetes, patients requiring hemodialysis
* Hypersensitivity to thalidomide, lenalidomide, or dexamethasone
* Previous therapy with pomalidomide
* Peripheral neuropathy ≥ Grade 2
* Incidence of gastrointestinal disease that may significantly alter the absorption of pomalidomide
* Subjects who received any of the following within the last 14 days of initiation of study treatment: plasmapheresis, major surgery, radiation therapy, or use of any anti-myeloma drug therapy
* Use of any investigational drugs within 28 days prior to enrollment
* Subjects with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis, and lupus, etc.
* Patients unable or unwilling to undergo antithrombotic prophylactic treatment
* Subjects who received an allogeneic hematopoietic stem cell transplant less than 12 months prior to enrollment
* Subjects who are planning for or eligible for hematopoietic stem cell transplant
* Pregnant or lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 2 years

SECONDARY OUTCOMES:
Progression-free Survival | up to 2 years
Duration of Response | up to 2 years
Time to Response | up to 2 years
Overall Survival | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MD, Principal Investigator — Blood Diseases Hospital Chinese Academy of Medical Sciences
Locations (1):
- Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided